CLINICAL TRIAL: NCT07101354
Title: A Phase I/Ⅱa, Single-arm, Open-label Trial of DGPR1008 for Intraoperative Fluorescence Imaging of Prostate-specific Membrane Antigen-positive Prostate Cancer
Brief Title: Research on PSMA-Targeted Intraoperative Fluorescent Imaging Agents
Acronym: DGPR1008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haitao Niu, MD (Other)
Responsible Party: Sponsor-Investigator, Haitao Niu, MD, Clinical Professor, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: QYFYEC2024-047-01; CXHL2400243 (Other: NMPA)
Record Dates: First submitted 2025-05-18; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer Patients Undergoing Radical Prostatectomy; Prostate CA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0.01mg/kg DGPR1008 Injection Dose Group 1 (n=6) (Experimental): On the day of administration, subjects will be randomized to receive the DGPR1008 Injection (0.01 mg/kg; n=6) via slow IV infusion over 60-90 minutes.
  Infusion Monitoring: Closely assess for infusion reactions; discontinue if necessary.
  Post-Infusion: Inspect injection site for erythema, pruritus, etc. Protocol Adherence: Conduct bio-sample collection, safety checks, and document all adverse events/concomitant therapies.
  Interventions: Drug: 0.01mg/kg DGPR1008 Injection Dose Group 1 (n=6)
- 0.02mg/kg DGPR1008 Injection Dose Group 2 (n=6) (Experimental): On the day of administration, subjects will be randomized to receive the investigational product (0.02 mg/kg; n=6) via slow IV infusion over 60-90 minutes.
  Infusion Monitoring: Closely assess for infusion reactions; discontinue if necessary.
  Post-Infusion: Inspect injection site for erythema, pruritus, etc. Protocol Adherence: Conduct bio-sample collection, safety checks, and document all adverse events/concomitant therapies.
  Interventions: Drug: 0.02mg/kg DGPR1008 Injection Dose Group 2 (n=6)
- Dose Group 0 (n=8) (Placebo Comparator): On the day of administration, subjects will be randomized to receive placebo (n=8) via slow IV infusion over 60-90 minutes.
  Infusion Monitoring: Closely assess for infusion reactions; discontinue if necessary.
  Post-Infusion: Inspect injection site for erythema, pruritus, etc. Protocol Adherence: Conduct bio-sample collection, safety checks, and document all adverse events/concomitant therapies.
  Interventions: Drug: Dose Group 0 (n=8)
- 0.04mg/kg DGPR1008 Injection Dose Group 3 (n=6) (Active Comparator): On the day of administration, subjects will be randomized to receive the investigational product (0.04 mg/kg; n=6) via slow IV infusion over 60-90 minutes.
  Infusion Monitoring: Closely assess for infusion reactions; discontinue if necessary.
  Post-Infusion: Inspect injection site for erythema, pruritus, etc. Protocol Adherence: Conduct bio-sample collection, safety checks, and document all adverse events/concomitant therapies.
  Interventions: Drug: 0.04mg/kg DGPR1008 Injection Dose Group 3 (n=6)
- 0.08mg/kg DGPR1008 Injection Dose Group 4 (n=6) (Active Comparator): On the day of administration, subjects will be randomized to receive the DGPR1008 Injection (0.08 mg/kg; n=6) via slow IV infusion over 60-90 minutes.
  Infusion Monitoring: Closely assess for infusion reactions; discontinue if necessary.
  Post-Infusion: Inspect injection site for erythema, pruritus, etc. Protocol Adherence: Conduct bio-sample collection, safety checks, and document all adverse events/concomitant therapies.
  Interventions: Drug: 0.08mg/kg DGPR1008 Injection Dose Group 4 (n=6)

INTERVENTIONS:
Drug: 0.01mg/kg DGPR1008 Injection Dose Group 1 (n=6) — Within the specified time period, conduct dose escalation, and administer the corresponding dose via intravenous drip according to the randomization information.
  Other Names: DGPR1008; 0.01mg/kg Dose Group 1 (n=6)
  Arms: 0.01mg/kg DGPR1008 Injection Dose Group 1 (n=6)
Drug: 0.02mg/kg DGPR1008 Injection Dose Group 2 (n=6) — Within the specified time period, conduct dose escalation, and administer the corresponding dose via intravenous drip according to the randomization information.
  Other Names: 0.02mg/kg Dose Group 2 (n=6); DGPR1008; Treatment group
  Arms: 0.02mg/kg DGPR1008 Injection Dose Group 2 (n=6)
Drug: 0.04mg/kg DGPR1008 Injection Dose Group 3 (n=6) — Within the specified time period, conduct dose escalation, and administer the corresponding dose via intravenous drip according to the randomization information.
  Other Names: 0.04mg/kg Dose Group 3 (n=6); DGPR1008; Treatment group
  Arms: 0.04mg/kg DGPR1008 Injection Dose Group 3 (n=6)
Drug: 0.08mg/kg DGPR1008 Injection Dose Group 4 (n=6) — Within the specified time period, conduct dose escalation, and administer the corresponding dose via intravenous drip according to the randomization information.
  Other Names: DGPR1008; 0.08mg/kg Dose Group 4 (n=6); Treatment group
  Arms: 0.08mg/kg DGPR1008 Injection Dose Group 4 (n=6)
Drug: Dose Group 0 (n=8) — Within the specified time frame, dose escalation will be conducted. Intravenous infusions will be administered according to randomization, with subjects receiving either the corresponding dose or placebo.
  Other Names: placebo control group
  Arms: Dose Group 0 (n=8)

SUMMARY:
Phase I:

Primary Research Objective:

Evaluate the safety, tolerability, and pharmacokinetic characteristics of a single dose of DGPR1008 in healthy subjects.

Secondary Research Objective:

Based on the safety and pharmacokinetic results, assess the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of DGPR1008.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent prior to the trial, and fully understand the trial content, procedures, and potential adverse reactions.
* Be able to complete the study as required by the trial protocol.
* Be an adult male aged 18-65 years (inclusive).
* Have a body weight ≥50 kg and a body mass index (BMI) of 18-30 kg/m² (calculated as BMI = weight [kg]/height² [m²]).
* Neither the subject nor their partner/spouse plan to conceive or donate sperm from screening until 3 months after the trial completion, and agree to use effective non-pharmacological contraception during the study.

Exclusion Criteria:

Subjects will be excluded if any of the following apply:

* Clinically significant abnormalities (physical exam, vital signs, ECG, labs) or severe medical history (cardiac, hepatic, renal, GI, neurological, respiratory, psychiatric, metabolic) deemed unsuitable by the investigator.
* History of allergy (≥2 drugs/foods, milk/pollen), or allergy to investigational drug/components.
* Alcohol abuse (>14 units/week) in prior 3 months or positive breathalyzer.
* Positive serology for HBsAg, anti-HCV, anti-HIV, or syphilis.
* Positive urine drug screen, drug abuse history (past 5 years), or illicit drug use (past 3 months).
* Blood loss >400 mL or platelet donation (2 therapeutic units) in prior 3/1 months, respectively.
* Smoking >5 cigarettes/day (past 3 months) and inability to abstain.
* Surgery within prior 3 months.
* Participation in another clinical trial (investigational product) within prior 3 months.
* Prescription medication use within prior 1 month.
* OTC drugs, herbal supplements, or vitamins within prior 48 hours.
* Other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 5 Days
  Incidence of Treatment-Emergent Adverse Events
Number of participants with abnormal vital signs | through study completion, an average of 5 Days
  temperature in ℃
Number of participants with abnormal vital signs | through study completion, an average of 5 Days
  pulse in beats/minute
Number of participants with abnormal vital signs | through study completion, an average of 5 Days
  blood pressure in mmHg
The number of participants with abnormal BMI | through study completion, an average of 5 Days
  Weight and height will be combined to report BMI in kg/m^2
Number pf participants with abnormal laboratory tests results | through study completion, an average of 5 Days
  complete blood count
Number pf participants with abnormal laboratory tests results | through study completion, an average of 5 Days
  blood chemistry panel
Number pf participants with abnormal laboratory tests results | through study completion, an average of 5 Days
  urinalysis

SECONDARY OUTCOMES:
Evaluation indices for pharmacokinetics(Cmax) | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  Cmax
Evaluation indices for pharmacokinetics(AUC(0-t)) | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  AUC(0-t)
Evaluation indices for pharmacokinetics(AUC(0-∞)) | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  AUC(0-∞)
Evaluation indices for pharmacokinetics(AUC_%Extrap) | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  AUC_%Extrap
Evaluation indices for pharmacokinetics(t1/2) | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  t1/2
Evaluation indices for pharmacokinetics(CL) | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  CL
Evaluation indices for pharmacokinetics(CLRenal) | PK Urine Samples:Pre-dose (within 120 minutes before dosing); During dosing (from start to end of infusion), Post-dose time intervals: 0-2hours, 2-4hours, 4-8hours, 8-12hours, 12-24hours, 24-48 hours.
  CLRenal
Evaluation indices for pharmacokinetics | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  λz
Evaluation indices for pharmacokinetics(Vz) | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  Vz
Evaluation indices for pharmacokinetics（MRT(0-t)、MRT(0-∞)） | PK Blood Samples:Pre-dose (within 60 minutes before dosing);Immediately after dosing completion (within 2 minutes),5 minutes(±2 minutes) and 15minutes (±3 minutes) and 30minutes (±5 minutes) and(1, 2, 4, 6, 8, 24 hours)(±30 minutes) post-dose.
  （MRT(0-t)、MRT(0-∞)）

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF